CLINICAL TRIAL: NCT02079324
Title: A Single Center, Open-Label, Accelerated Titration, Dose-Escalating, Phase Ι Study to Evaluate the Safety and Tolerability of IT Injection GX-051, Stem Cell Based Gene Therapeutics in Patients With Very Advanced Head and Neck Cancer
Brief Title: Genetically Modified Mesenchymal Stem Cell Theraopeutic Against Head and Neck Cancer
Acronym: GX-051
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Genexine, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GX-051_HNC_1
Record Dates: First submitted 2014-02-27; First posted 2014-03-05 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2014-03

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; gene therapy; stem cell therapy; immunotherappy
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GX-051 (Experimental): GX-051 intratumoral injection
  Interventions: Biological: GX-051

INTERVENTIONS:
Biological: GX-051 — intratumoral injection

SUMMARY:
The purpose of this research is to evaluate MTD, Safety and efficacy of GX-051 after intratumoral injection in head and neck cancer patience.

DETAILED DESCRIPTION:
The primary purpose of the study is to determine MTD(Maximum Tolerable Dose) of GX-051 administered in tumor. The second purpose is to evaluate safety and efficacy of GX-051.

ELIGIBILITY:
Inclusion Criteria:

* Are capable of understanding and complying with the requirements of the study and have signed the informed consent from (ICF).
* Very advanced head and neck cancer aged more than 19.
* Longest distance of the tumor is bigger than 1 cm and capable of Intratumoral injection.
* Baseline ECOG Performance Status 0, 1 or 2.
* Have a life expectancy more than 6 months.

Exclusion Criteria:

* Have no history of prior anticancer treatment.
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.Subject who have participated in a clinical trial of an treatment vaccine or immunotherapy in an year.
* Have a tumor which is near a main vessel that can be occured embolism after injection or which has hypervascularity.
* Patients currently receiving anticancer immuno-therapies Patients who have received prior treatment with an stem cell therapy.
* Have autoimmune disease (multiple sclerosis, systemic lupus erythromatosis, thyroiditis, psoriasis, inflammatory bowel diseases etc.).
* Have Graft rejection reaction such as GVHD.
* Have immunodeficiency disease.
* Leukocytes< 3.0 x109/L.
* Absolute neutrophil count < 1.5x109/L.
* Platelet count < 100 x 109/L.
* Have known positive test for hepatitis B surface antigen, hepatitis C antibody, and human immunodeficiency virus (HIV).
* Alanine Aminotransferase (ALT) > 2.5xUNL.
* Aspartate Aminotransferase (AST)> 2.5xUNL.
* Total Bilirubin> UNL.
* Have blood Creatinine> UNL.
* Known allergy to IL-12 or the excipient(s) of the study medication including fetal bovine serum.
* Second primary cancer Metastatic brain tumor or meningioma.
* Have a tumor near a main artery.
* Uncontrolled hypertension.
* Uncontrolled diabetes uncontrolled (arrhythmia).
* Heart failure (more than NYHA Functional Class II); unstable coronary artery disease; myocardial infarction within 6 months.
* Child-Pugh Class C hepatic impairment.
* Severe renal impairment (creatinine clearance < 30 ml/min) or on dialysis.
* Have active infection or history of recurrent infection.
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study.
* Are considered ineligible by the investigator due to a mental disease or CNS disease.
* Administration of any other tumor therapy, including chemotherapy and radiotherapy within 4 weeks(6 weeks in case of nitrosoureas and mytomycin C) before the beginning of study treatment.
* Patients receiving chronic, systemic treatment with immunosuppressive agent(steroid) or immuno-modulator within 2 weeks prior to screening.
* Have participated in another clinical trial within 30 days prior to dosing.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2014-03; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
MTD after GX-051 intratumoral injection | 2 months

SECONDARY OUTCOMES:
Adverse events after GX-051 intratumoral injection | 2 months
Anti-tumor response by RECIST 1.1 on computed tomography | 2 months
  Response Evaluation Criteria in Solid Tumors (RECIST) are used to determine objective clinical response. Complete Rresponse (CR) is the disappearance of all target lesions, partial response (PR) is at least a 30% decrease in the target lesions, progressive disease (PD) is at least a 20% increase in the target lesions or appearance of one or more new lesions, and stable disease (SD) is neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD.
Changes of INF-γ and IL-12 levels in blood comparing to the baseline after GX-051 intratumoral injection | 2 months
  unit: pg/ml
Changes of immune cell distribution in tumor tissue after GX-051 intratumoral injection | 2 months
  We will analyze immune cells such as CD4+ T cell, CD8+ T cell, NK cell by FACS analysis on day 1(baseline), day 29(end of treatment) and day 57(follow up)
Evaluation of antibody generation against IL-12 which is active ingredient of GX-051 | 2 months
  We will analyze anti-IL-12 antibody in blood by ELISA on the screening visit and the follw up visit. Result will report as existence or absence of the anti-body .
Evaluation of long term safety examined by vital sign, physical examination, clinical laboratory tests, CT etc | 17 monthes
  Safety profile would be examined by vital sign, physical examination, clinical laboratory tests, CT etc

CONTACTS AND LOCATIONS:
Overall Officials: Minsik Kim, M.D., Principal Investigator — Seoul St.Mary's Hospital of the Catholic University of Korea; Hyun-Tak Jin, ph.D., Study Director — Genexine, Inc.
Locations (1):
- Seoul St.Mary's Hospital of the Catholic University of Korea, Seoul, South Korea